CLINICAL TRIAL: NCT00518388
Title: Perceptions of Cervical Cancer and Human Papillomavirus Among Asian Americans
Brief Title: Perceptions of Cervical Cancer Among Asian Americans
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2007-0101
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Epidemiology
Keywords: Epidemiology; Cervical Cancer; Human Papillomavirus; Focus Group; Questionnaire; Survey; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focus Group + Questionnaire: Participants that are self identified as Korean, Filipino, or Vietnamese.
  Interventions: Behavioral: Focus Group; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Focus Group — Focus groups each lasting about 2 hours.
Behavioral: Questionnaire — Questionnaire relating to your health practices and knowledge about cervical cancer and HPV.
  Other Names: Survey

SUMMARY:
The goal of this research study is to learn about the beliefs, practices, and knowledge about cervical cancer among Asian American young adults. Researchers want to develop materials that will educate Asian Americans about cervical cancer and encourage them to get screened for this disease.

DETAILED DESCRIPTION:
Survey:

If you agree to take part in this study, you will complete a survey about your health practices and knowledge about cervical cancer and HPV. You will also be asked to provide some personal history on yourself such as your age, gender, birthplace, ethnicity, relationship status and educational level. Female participants will be asked to indicate if they have received an HPV test (also called a "Pap" test) within the last 3 years. The survey will take about 5-10 minutes to complete and will be filled out on the same day as the focus group.

Focus Group:

You will also take part in a discussion group called a "focus group." A trained focus group leader will guide you and 8-10 others through a series of questions. He/she will lead a discussion to hear comments, opinions, and observations on a brochure and poster about cervical cancer and HPV. Groups will be made up of participants of the same gender (that is, all male or all female) and ethnic group (Filipino, Korean, or Vietnamese). Each discussion group will last about 2 hours and may be audiotaped so that the discussion may be transcribed and analyzed. You will only be called by your first name and you are not required to use your real name during the focus group discussion. You will not be identified by the audiotape recordings.

Length of Study:

When the focus group discussion is over, you will be off-study.

This is an investigational study. Up to 60 participants will be enrolled on this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Self identified as Korean, Filipino, or Vietnamese
2. Individuals 18-29 years of age
3. Have a high school education or less (but not less than 4th grade)
4. Able to read and speak English and one of these languages: Korean, Vietnamese, or Tagalog
5. Lower socioeconomic status, defined as: for a household of 1, not more than $18,620 annual income, for a household of 2, not more than $24,980, for a household of 3, not more than $31,340, for a household of 4, not more than $37,700, for a household of 5, not more than $44,060, for a household of 6,not more than $50,420, for a household of 7, not more than $56,780 NOTE: The CDC has granted some flexibility with these income guidelines
6. Not currently pregnant

Exclusion Criteria:

1) Household income greater than 200% of the federal poverty level

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants that are self identified as Korean, Filipino, or Vietnamese.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To learn about the beliefs, practices, and knowledge about cervical cancer among Asian American young adults | 1 Year

SECONDARY OUTCOMES:
To develop materials that will educate Asian Americans about cervical cancer and encourage them to get screened for this disease | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Hajek, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org